CLINICAL TRIAL: NCT03071094
Title: A Phase I/IIa Trial to Evaluate the Safety and Efficacy of the Combination of the Oncolytic Immunotherapy Pexa-Vec With the PD-1 Receptor Blocking Antibody Nivolumab in the First-line Treatment of Advanced Hepatocellular Carcinoma (HCC)
Brief Title: A Trial to Evaluate the Safety and Efficacy of the Combination of the Oncolytic Immunotherapy Pexa-Vec With the PD-1 Receptor Blocking Antibody Nivolumab in the First-line Treatment of Advanced Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The decision was taken to stop prematurely the trial due to the failure of Pexa-Vec and nivolumab in their respective pivotal trials (i.e., PHOCUS and CheckMate 459).
Sponsor: Transgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG6006.01
Record Dates: First submitted 2017-02-10; First posted 2017-03-06 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pexa-Vec combined with Nivolumab - Phase I (Experimental): Participants were administered Pexa-Vec (pexastimogene devacirepvec) as 3 bi-weekly intratumoral (IT) injections of 10^9 pfu at day 1 and weeks 2 and 4 and nivolumab intravenously every 2 weeks (from week 2).
  Interventions: Biological: Pexastimogene Devacirepvec (Pexa Vec); Drug: Nivolumab
- Pexa-Vec combined with Nivolumab - Phase IIa (Experimental): Participants were administered Pexa-Vec (pexastimogene devacirepvec) as 3 bi-weekly intratumoral (IT) injections of 10^9 pfu at day 1 and weeks 2 and 4 and nivolumab intravenously every 2 weeks (from week 2).
  Interventions: Biological: Pexastimogene Devacirepvec (Pexa Vec); Drug: Nivolumab

INTERVENTIONS:
Biological: Pexastimogene Devacirepvec (Pexa Vec) — Pexa-Vec (pexastimogene devacirepvec) will be administered as 3 bi-weekly intratumoral (IT) injections of 10^9 pfu at day 1 and weeks 2 and 4
Drug: Nivolumab — Nivolumab will be administered intravenously every 2 weeks (from week 2)

SUMMARY:
This is a study to Evaluate the Safety and Efficacy of the Combination of the Oncolytic Immunotherapy Pexa-Vec With the PD-1 Receptor Blocking Antibody Nivolumab in the First-line Treatment of Advanced Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis of primary HCC, excluding cholangiocarcinoma, hepatocholangiocarcinoma, fibrolamellar carcinoma and hepatoblastoma
* Advanced stage HCC per EASL-EORTC (European Association for the Study of the Liver-European Organisation for Research and Treatment of Cancer) guidelines, i.e. patients who are not candidates for curative interventions and not candidates for locoregional modalities
* Patients naïve to systemic therapy for HCC
* Tumor status (as determined by radiology evaluation): At least one measurable viable tumor in the liver, ≥1 cm longest diameter (LD), using a dynamic imaging technique (arterial phase of triphasic computerized tomography [CT] scan, or dynamic contrast-enhanced magnetic resonance imaging [MRI]), and injectable under imaging-guidance (CT or ultrasound)
* At least one tumor that has not received prior local-regional treatment, or that has exhibited definitive growth of viable tumor since prior local-regional treatment of HCC undertaken at least 4 weeks prior to enrolment or 3 months prior to enrolment for radioembolization
* Child-Pugh Class A. Note: paracentesis, albumin infusion or diuretic treatment cannot be used to downgrade Child-Pugh score (e.g., to improve from severe to moderate/mild or from moderate to mild ascites)
* Performance status 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Adequate hematological, hepatic, and renal function
* Additional inclusion criteria exist

Exclusion Criteria:

* Histological diagnosis of cholangiocarcinoma, hepatocholangiocarcinoma, fibrolamellar carcinoma and hepatoblastoma
* Symptomatic cardiovascular disease, including but not limited to significant coronary artery disease (e.g., requiring angioplasty or stenting) or congestive heart failure within the preceding 12 months
* Current or past history of cardiovascular disease (e.g., past history of myocardial infarction, ischemic cardiomyopathy) unless cardiology consultation and clearance has been obtained for study participation
* History of moderate or severe ascites, bleeding esophageal varices, hepatic encephalopathy or pleural effusions related to liver insufficiency within 6 months of screening; patients with adequately treated esophageal varices are allowed
* Active, known or suspected significant immunodeficiency due to underlying illness including HIV/AIDS, autoimmune diseases, and/or immune-suppressive medication including high-dose corticosteroids
* History of severe eczema and/or ongoing severe inflammatory skin condition (as determined by the Investigator) requiring medical treatment
* Any known allergy or reaction to any component of nivolumab formulation or its excipients
* Additional exclusion criteria exist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Site No 0102, Nancy
  - Site No 0101, Paris

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant signed informed consent on 04 July 2017. Last participant last visit occurred on 03 February 2021.
Pre-assignment Details: Of 14 screened participants, 12 met eligibility criteria and were included in the trial. This was a Phase I/IIa trial with Phase I: single cohort of 6 patients assessing the safety of standard Pexa-Vec and nivolumab doses and Phase IIa: extension of the Phase I to up to 30 patients, assessing the efficacy and safety of Pexa-Vec and nivolumab. The trial was terminated prematurely during the Phase IIa due to the failure of Pexa-Vec and nivolumab in their respective pivotal trials in HCC.
Period: Overall Study
Arm/Group | Pexa-Vec Combined With Nivolumab - Phase I | Pexa-Vec Combined With Nivolumab - Phase IIa
Started | 7 | 5
Completed | 5 | 4
Not Completed | 2 | 1
Not completed — Death | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Phase I and Phase IIa: Participants who received at least one dose of either study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pexa-Vec Combined With Nivolumab - Phase I | Pexa-Vec Combined With Nivolumab - Phase IIa | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.1) | 62.8 (18.0) | 65.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9
Stage of HCC per BCLC (Barcelona Clinic Liver Cancer) [Count of Participants; unit: Participants] — As per the BCLC (Barcelona Clinic Liver Cancer) scale, the liver cancer stages range from stage 0 (less advanced stage of liver cancer) to stage D (more advanced stage of liver cancer):
  * Stage 0: very early stage of liver cancer, single nodule <2cm
  * Stage A: early stage of liver cancer, single nodule <5cm or up to 3 nodules <3cm
  * Stage B: intermediate stage of liver cancer, large multinodular
  * Stage C: advanced stage of liver cancer, portal invasion / extrahepatic spread
  * Stage D: terminal stage of liver cancer.
  Participants
    Stage 0 | 0 | 0 | 0
    Stage A | 0 | 0 | 0
    Stage B | 0 | 0 | 0
    Stage C | 7 | 5 | 12
    Stage D | 0 | 0 | 0
ECOG (Eastern Cooperative Oncology Group) performance status [Count of Participants; unit: Participants] — As per the ECOG (Eastern Cooperative Oncology Group) scale, the performance status is ranked from grade 0 (best performance status) to grade 4 (worst performance status) as follows:
  * Grade 0: fully active
  * Grade 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  * Grade 2: ambulatory and capable of all selfcare but unable to carry out any work activities
  * Grade 3: capable of only limited selfcare
  * Grade 4: completely disabled.
  Participants
    0 | 4 | 5 | 9
    1 | 3 | 0 | 3
    2 | 0 | 0 | 0
    3 | 0 | 0 | 0
    4 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs are occurrence of any following AE related to study drugs occurring during 4 weeks after 1st Pexa-Vec injection:
  1. Grade 3-4 non-hematologic toxicity representing a 2-grade increase over baseline, excluding: nausea, vomiting, diarrhea, fever>40.0°C lasting less than 24h (grade 3), alopecia, grade 3 fatigue* and grade 3 laboratory/metabolic abnormalities* (*returning to grade 2 or less within 72h)
  2. Grade ≥ 3 acute immune-related AE involving major organs
  3. Grade ≥ 3 injection site reaction
  4. AST or ALT ≥ 10xULN unless related to liver metastases progression; AST or ALT doubling concurrent with total bilirubin doubling
  5. Any toxicity resulting in treatment delay of 2 or more weeks
  6. Grade ≥ 3 or ≥ 2-grade neutropenia increase over baseline lasting >7 days, neutropenic fever, grade 4 thrombocytopenia (or grade 3 with bleeding)
  7. Association of LVEF less than LLN, blood troponin T or I increase above ULN and any ECG abnormality indicating grade 3 cardiac disorder.
Time Frame: 4 weeks from the first study drug administration
Population: Participants who received at least one dose of either study drug (excluding one patient who did not complete the 4 week-period from the first study drug administration).
Measure: Count of Participants; unit: Participants
Arm/Group | Pexa-Vec Combined With Nivolumab - Phase I
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Phase I: Number of Participants With Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence or effect in a patient, whether or not considered related to the protocol treatment, that at any dose: (i) results in death, (ii) is life-threatening, (iii) requires inpatient's hospitalization or prolongation of existing inpatients´ hospitalization, (iv) results in persistent or significant disability or incapacity, (v) is a congenital anomaly or birth defect, (vi) results in any other medically important condition.
Time Frame: 4 weeks from the first study drug administration
Population: Participants who received at least one dose of either study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pexa-Vec Combined With Nivolumab - Phase I
Number analyzed (Participants) | 7
Participants | 6

3. Primary Outcome: Overall Response Rate (ORR) According to RECIST 1.1.
Description: Overall Response Rate (ORR): proportion of patients, whose best overall response is either complete response (CR) or partial response (PR), confirmed at least 4 weeks after initial documentation.
Time Frame: 6 months from the first study drug administration
Population: The overall response rate (ORR) was calculated on the total number of participants included in Phase I and Phase IIa who received at least one dose of either study drug. Phase I and IIa patients did not differ in terms of eligibility criteria and study treatment and represented a total of 12 patients. Thus a single analysis of the ORR on the phase I/IIa sample size is more relevant than two separate analyses on very low sample sizes.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pexa-Vec Combined With Nivolumab - Phase I and Phase IIa: Participants were administered Pexa-Vec (pexastimogene devacirepvec) as 3 bi-weekly intratumoral (IT) injections of 10^9 pfu at day 1 and weeks 2 and 4 and nivolumab intravenously every 2 weeks (from week 2).
Arm/Group | Pexa-Vec Combined With Nivolumab - Phase I and Phase IIa
Number analyzed (Participants) | 12
Percentage of participants | 33.3 [9.9 to 65.1]

ADVERSE EVENTS:
Time Frame: Adverse events (and serious adverse events) were recorded from the first study drug administration up to 28 days after the last study drug dose.
Description: Adverse event information was collected by regular investigator assessment and regular laboratory testing.
Arm/Group | Pexa-Vec Combined With Nivolumab - Phase I | Pexa-Vec Combined With Nivolumab - Phase IIa
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/5
Serious Adverse Events (participants affected / at risk) | 6/7 | 4/5
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pexa-Vec Combined With Nivolumab - Phase I (N=7) | Pexa-Vec Combined With Nivolumab - Phase IIa (N=5)
Pyrexia (General disorders) | 2 (3) | 0 (0)
Influenza Like Illness (General disorders) | 1 (2) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (6) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tumour Necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pexa-Vec Combined With Nivolumab - Phase I (N=7) | Pexa-Vec Combined With Nivolumab - Phase IIa (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (3)
Ascites (Gastrointestinal disorders) | 2 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (3) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (4)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 5 (6)
Chills (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (4) | 0 (0)
Influenza like illness (General disorders) | 1 (3) | 3 (5)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 5 (6) | 0 (0)
Pyrexia (General disorders) | 7 (16) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0)
Rash pustular (Infections and infestations) | 3 (3) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
C-reactive protein (Investigations) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Strangury (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (7) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (6) | 2 (8)
Hypotension (Vascular disorders) | 2 (5) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely as per Sponsor's decision based on the failure of Pexa-Vec and nivolumab in their respective pivotal trials in HCC. As a consequence, the enrollment in Phase IIa was not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT03071094/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03071094/SAP_001.pdf